CLINICAL TRIAL: NCT04266119
Title: Online HOPE Intervention on Mental Health Literacy Among Youths in Singapore: An RCT Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Piyanee KLAININ-YOBAS, Associate Professor from National University of Singapore (Unknown); Yong Shian Shawn GOH, Assistant Professor from National University of Singapore (Unknown)
Responsible Party: Principal Investigator, Tay Jing Ling, Graduate Student, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S-19-251; NYF/Jul19/01 (Other Grant/Funding Number: National Youth Fund)
Record Dates: First submitted 2020-02-06; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Mental Health Literacy; Depression Literacy; Psychological Well-being; Stress, Psychological
MeSH Terms: conditions — Psychological Well-Being; Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The HOPE intervention can be accessed through web. It consists of two sessions per week, with a total of four sessions. In this study, participants will be sent weekly weblinks for access to each session. Each session take about ten minutes to complete. Each session consist of pre-post multiple-choice and/or open-end question, video(s) and mental health information. The first session is about depression. The second session is about positive psychology and consists of relevant exercises such as gratitude, affect-based and strength-based exercises. The third session describes anxiety disorder. The last session describes relaxation techniques and self-management of unhelpful thoughts.
  Each session consists of quizzes, video(s), and graphical / written information
  Interventions: Behavioral: Online HOPE intervention
- Control (Active Comparator): The group will receive a control website intervention that consists of several graphical inspirational quotes. Examples of the quotes are, 'Today is full of possible' and 'You can do anything'.
  Interventions: Behavioral: Online HOPE intervention

INTERVENTIONS:
Behavioral: Online HOPE intervention — Online HOPE intervention to increase mental health literacy

SUMMARY:
The author developed the HOPE intervention based on a systematic review (Tay, Tay, & Klainin-Yobas, 2018). The overall aim of the study is to test the effectiveness of the online HOPE intervention in enhancing mental health literacy, depression literacy, psychological well-being and in reducing stress among youths aged 18 - 24 living in Singapore.

DETAILED DESCRIPTION:
The study will be a two-group, parallel randomized control trial (RCT), with a pre-test, post-test and repeated, control group design.

he overall aim of the study is to test the effectiveness of the online HOPE intervention in enhancing mental health literacy, on depression literacy, psychological well-being and in reducing stress among youths aged 18 - 24 living in Singapore.

ELIGIBILITY:
Inclusion Criteria:

* : a) students of a particular University in Singapore, b) aged between 18 to 24 years old, c) had internet access and d) could read, write and understand the English language.

Exclusion Criteria:

* Exclusion criteria were reading or hearing disabilities. This was because the online HOPE intervention consists of written words and videos that require visual and auditory abilities, respectively.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Depression Literacy | Change from baseline depression literacy to post intervention (up to 1 month), and follow up at 2 months
  using D-Lit. The scale consists of 22 items that are scored 'true', 'false' or 'don't know'. Greater scores equate greater depression MHL.
Anxiety literacy | Change from baseline depression literacy to post intervention (up to 1 month), and follow up at 2 months
  A-Lit. The scale consists of 22 items that are scored 'true', 'false' or 'don't know'. Greater scores equate greater anxiety MHL.
Mental health literacy | Change from baseline depression literacy to post intervention (up to 1 month), and follow up at 2 months
  depression vignette (shortened)

SECONDARY OUTCOMES:
Psychological well-being | Change from baseline depression literacy to post intervention (up to 1 month), and follow up at 2 months
  Ryff's Psychological Well-Being Scale. PWB can be measured by the 18-items psychological well-being scale that measures the six dimensions of PWB (Ryff, 1989). The scale ranges from 1 (strongly disagree) to 7 (strongly agree). Scores ranged from 18 to 123, with greater points indicating greater PWB.
Stress | Change from baseline depression literacy to post intervention (up to 1 month), and follow up at 2 months
  Perceived Stress Scale. The 10-question perceived stress scale (PSS) consists of five response categories: never (0), almost never (1), sometimes (2), fairly often (3), and very often (4). Total scores range from 0 to 56, with higher scores indicating higher stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ling Tay, MN, Principal Investigator — Singapore University of Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tay JL. Online HOPE intervention on help-seeking attitudes and intentions among young adults in Singapore: A randomized controlled trial and process evaluation. Arch Psychiatr Nurs. 2022 Dec;41:286-294. doi: 10.1016/j.apnu.2022.09.008. Epub 2022 Sep 17. PMID 36428062
- [Derived] Tay JL, Goh YSS, Sim K, Klainin-Yobas P. Impact of the HOPE Intervention on Mental Health Literacy, Psychological Well-Being and Stress Levels amongst University Undergraduates: A Randomised Controlled Trial. Int J Environ Res Public Health. 2022 Aug 8;19(15):9772. doi: 10.3390/ijerph19159772. PMID 35955126